CLINICAL TRIAL: NCT03582670
Title: Prospective Memory Training in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201709182
Record Dates: First submitted 2018-06-06; First posted 2018-07-11 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
Keywords: Prospective Memory; Occupational Therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strategy Training Intervention (Experimental): Study participants receive specific memory strategy training with training games, as well as feedback on accuracy and performance.
  Interventions: Behavioral: Strategy Training
- Process Training (Active Comparator): Study participants attend training sessions and complete training games, but receive no specific strategy training
  Interventions: Behavioral: Process Training
- Control Group (Other): Study participants do not attend any strategy training sessions.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Strategy Training — Participants will attend four strategy training sessions total. In sessions 1 and 2, in addition to teaching about event- and time-based tasks, the trainer teaches the participant specific strategies for each type of task (implementation intentions for event-based and strategic clock-checking for time-based). In sessions 3 and 4, the trainer tells the participant s/he will be practicing both types of tasks in the training games and can support the participant's strategy use if needed. Feedback on accuracy and strategy use are provided after each training game. At the end of each session after completing the training games, the trainer and participant discuss how the strategies can be applied to the participant's real-life prospective memory goals, and the trainer helps the participant develop written action plans to do so. Plans are reviewed (and modified if necessary) at each session.
  Arms: Strategy Training Intervention
Behavioral: Process Training — Participants will attend four process training sessions in this group. In sessions 1 and 2, the trainer teaches the participant about event- and time-based prospective memory tasks, respectively. In sessions 3 and 4, the trainer simply tells the participant that s/he will be practicing both types of tasks in the training games. In all sessions, the participant completes the training games with no strategy instruction from the trainer. Feedback on accuracy is provided after each training game. At the end of each session after completing both training games, the trainer reminds the participant of his/her real-life prospective memory goals, provides a handout that lists the goals, and instructs the participant to try to complete them as intended. Of note, even this minimal level of discussion of real-life cognitive tasks is not typical of process training interventions, but we include it to control for that which is occurring in the strategy training group.
  Arms: Process Training
Behavioral: Control Group — Participants in this group do not attend any sessions during the time the other groups are participating in the Strategy or Process Training
  Arms: Control Group

SUMMARY:
The long term goal of this work is to reduce disability among people with Parkinson disease (PD) by enabling them to cope with cognitive decline so they can perform and participate in desired activities and roles. This project focuses on prospective memory, or the ability to remember to execute delayed intentions at the appropriate moment in the future. The current study tests the effects of two primary cognitive intervention approaches (process training & strategy training) on prospective memory performance in PD. The investigators will conduct a single-blind randomized controlled trial in which individuals with mild cognitive impairment in PD (PD-MCI; N = 90) will complete pre-training assessment, randomization to training group (control, process training, strategy training), four training sessions (process and strategy training groups), and post-training assessment.

DETAILED DESCRIPTION:
RANDOMIZATION

Once a participant is enrolled in the study and completes the Pre-testing session (described in detail below), they will be randomized into one of the following study groups:

1. Process Training Group - the trainer teaches the participant about event- and time-based prospective memory tasks, respectively. The trainer simply tells the participant that s/he will be practicing both types of tasks in training games.
2. Strategy Training Group - In training sessions 1 and 2, in addition to teaching about event- and time-based tasks, the trainer teaches the participant specific strategies for each type of task (implementation intentions for event-based and strategic clock-checking for time-based; and instructs in their use before and during the training games.
3. Contro1 Group - Receives no training sessions. Only Completes the PRE, POST and 1-month & 3-month Follow Up portions of the study.

STUDY VISITS

* On the day of their testing appointment, participants will arrive at their designated location at the WUSM Movement Disorders Clinic for their testing session. All participants will provide written informed consent before their first testing session begins, and the examiner will answer any questions before beginning testing. Scheduled participants will be mailed or emailed (depending on their preference) study information and a copy of the consent form. Participants will receive reminder calls 1-2 days before their appointments.
* Demographics will be collected on all participants. This includes age, gender, years of education, living status, race, and ethnicity after consent is obtained. This can be completed online via Redcap or on paper at the testing session.
* Investigators will collect PD clinical characteristics from the Movement Disorders Clinical Record. Clinical Characteristics includes: Hoehhn & Yahr Stage, year of first PD symptoms, year of initial PD diagnosis, MoCA score at most recent clinic visit, Side of symptom onset, type of symptom onset (tremor vs. bradykinesia), PD medications, and most recent Unified Parkinson Disease Rating Scale Motor Score.

Participant Questionnaires:

Participants will complete the PRMQ, CAPM, IPA and BDI questionnaires.

* Prospective and Retrospective Memory Questionnaire (PRMQ; attached) - Used to rate the participant's everyday retrospective and prospective memory.
* Comprehensive Assessment of Prospective Memory (CAPM; attached) - Used to rate the participant's everyday prospective memory
* Impact of Participation and Autonomy (IPA; attached)- A questionnaire about the participant's ability to take part in daily activities.
* Beck Depression Inventory (BDI, attached) - Used to characterize current depression, which is common in PD.

Informant Report Questionnaires:

Participant's will identify an informant (spouse, relative, or close friend) to fill out the PRMQ Proxy Report, a Self-Reported CAPM, and a CAPM - Proxy Report.

Demographics will be collected on all informants. This includes age, gender, years of education, living status, race, and ethnicity.

Participant and Informant questionnaires can be filled out prior to the study session via Redcap. Most participants request this method because it saves them time on the day of the study session. The online questionnaires have a consent form to look over before filling them out (see attached online consent), and the participant agrees to the consent by clicking "Next" in the online form, and completing the questionnaires; if participants elect to complete the questionnaires on paper, they can complete them at their testing session. The research team will will first go over the written consent with them at the session before the participant fills out the written questionnaires. Experimenters will check the questionnaires for completion. This procedure will also be followed if the participant elects to fill out the online questionnaire in Redcap.

Testing sessions:

Participants will perform testing while on their regular PD medications.

Pre-training Assessment: (1.5 hours) - MoCA and Virtual Week.

* The Montreal Cognitive Assessment (MoCA; attached) will be administered to assess global cognition at the time of the study visit.
* The Virtual Week test (attached) will be administered to the participant. It is a computerized board game that simulates daily life and real-world prospective memory challenges. Each circuit represents one day in which the participant completes time-appropriate activities and makes choices about them (i.e. the ongoing activity). Each day has 8 prospective memory tasks (4 event based, 4 time based). Participants complete a practice day and then three test days, with equivalent versions counterbalanced across Pre and Post testing. The main outcome variable is the proportion of correct prospective memory responses for each task type (12 event based, 12 time based).

Strategy Training Sessions (GROUPS 1-Process Training AND 2-Strategy Training ONLY): These are 4 sessions that occur over the next 2 weeks after the Pre-training Assessment. (1 HOUR EACH) GROUP 1, Process training: In sessions 1 and 2, the trainer teaches the participant about event- and time-based prospective memory tasks, respectively. In sessions 3 and 4, the trainer simply tells the participant that s/he will be practicing both types of tasks in the training games. In all sessions, the participant completes the training games with no strategy instruction from the trainer. Feedback on accuracy is provided after each training game. This is typical of a process training approach and expects that either practice of the training tasks will improve prospective memory ability per se or participants will develop effective strategies for completing prospective memory tasks on their own. At the end of each session after completing both training games, the trainer reminds the participant of his/her real-life prospective memory goals, provides a handout that lists the goals, and instructs the participant to try to complete them as intended. It should be noted that the inclusion of even this minimal level of discussion of real-life cognitive tasks is not typical of process training interventions.

GROUP 2, Strategy Training: In training sessions 1 and 2, in addition to teaching about event- and time-based tasks, the trainer teaches the participant specific strategies for each type of task (implementation intentions for event-based and strategic clock-checking for time-based) and instructs in their use before and during the training games. In sessions 3 and 4, the trainer tells the participant s/he will be practicing both types of tasks in the training games and can support the participant's strategy use if needed. Feedback on accuracy and strategy use are provided after each training game. At the end of each session after completing the training games, the trainer and participant discuss how the strategies can be applied to the participant's real-life prospective memory goals, and the trainer helps the participant develop written action plans to do so. Plans are reviewed (and modified if necessary) at each session.

* The Bangor Goal-Setting Interview (BGSI) - The BGSI is a structured assessment developed for use in cognitive rehabilitation research. It offers a standardized means of eliciting individual goals and rating goal attainment over time and has been successfully used in RCTs with older adults, including those with mild to moderate dementia. During the first two training sessions, after an explanation of the prospective memory task types (session 1: event, session 2: time), participants complete the BGSI with the trainer to identify and set goals for their real-life prospective memory tasks. Participants identify up to 6 prospective memory tasks they anticipate having to complete over the next 2 weeks (before Post assessment), define goals for completing each task, and describe what needs to happen for the goal to be considered partially (25%, 50%, and/or 75%) and fully achieved.
* Credibility/ Expectancy Questionnaire (CEQ; attached) - this will be completed by the participant after the second training session to rate how credible they think the strategy instruction training is, and how well they think it will work on 1) their performance on the computer task, and 2) their performance in everyday life.

Post-training Assessment (1.5 hours) - (For Groups 1 (Process) and 2 (Strategy) = One week after the last training session; For Group 3 (Control) = 3-4 weeks after the Pre-Training Assessment): Virtual Week and NIH Toolbox Cognitive Battery

* The Virtual Week Task will be administered again, but with new tasks to remember.
* The NIH Toolbox Cognitive Battery (instructions attached) will be administered to obtain an overall measure of executive function. This battery includes a Picture Vocabulary Test, Picture Sequence Memory Test, Flanker Inhibitory Control and Attention Test, Dimensional Change Card Sort Test, List Sorting Working Memory Test, Pattern Comparison, and Oral Reading Test.
* GROUPS 1 (Process) and 2 (STRATEGY) ONLY: Based on their BGSI interview during the training sessions, participants report on their performance of each task and, in collaboration with the trainer, rate each task for attainment on a 10-point scale using the previously determined descriptors as reference (higher scores indicate better goal attainment). Task attainment scores are averaged to yield a mean attainment score.

One-month Follow-up Assessment (40 minutes) (One month after the Post Training Assessment):

The PRMQ, IPA and CAPM Questionnaires will be given to participants for a second time as follow-up online in Redcap or by mail (depending on the participant's preference).

The study informant will fill out proxy-reported PRMQ and CAPM for a second time as a follow-up online in Redcap or by mail (depending on the informant's preference).

Three-month Follow-up Assessment (40 minutes) (Three months after the Post Assessment):

The PRMQ, CAPM, and IPA Questionnaire will be given to participants for a third time as follow-up online in Redcap or by mail (depending on the participant's preference).

The study informant will fill out proxy-reported PRMQ and CAPM for a third time as a follow-up online in Redcap or by mail (depending on the informant's preference).

ELIGIBILITY:
Inclusion Criteria:

* Males and females over age 50
* Meet criteria for typical idiopathic PD
* Hoehn & Yahr stage I-III
* Treated with levodopa/carbidopa
* Have PD with Mild Cognitive Impairment (PD-MCI) according to Movement Disorders Society (MDS) Level II diagnostic criteria.
* Medications should be stable for 4 weeks prior with no changes planned during the study (we will document any unplanned changes).

Exclusion Criteria:

* Dementia according to MDS criteria or MoCA score <21
* Other neurological disorders,
* Brain surgery
* History of psychotic disorder
* Change in medication during the study
* Treatment with medications that interfere with cognition (e.g. anticholinergics)
* Any condition that would interfere with participation (e.g., non-English speaking, significant current depression).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Virtual Week | 4 to 6 weeks
  A computerized board game that simulates daily life and real-world prospective memory challenges. Each circuit represents one day in which the participant completes time-appropriate activities and makes choices about them (i.e. the ongoing activity). Each day has 8 prospective memory tasks (4 event based, 4 time based). Participants complete a practice day and then three test days, with equivalent versions counterbalanced across Pre and Post testing. The main outcome variable is the proportion of correct prospective memory responses for each task type (12 event based, 12 time based). Change of performance on the Virtual Week from the Pre- and Post-session will be measured.
Prospective and Retrospective Memory Questionnaire | Through completion of the study, up to 16 weeks.
  Used to rate the participant's everyday retrospective and prospective memory. Change in scores on this questionnaire will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No